CLINICAL TRIAL: NCT06318559
Title: RIDERS: Artificial Intelligence 3D Augmented Reality Robot-Assisted-Radical- Prostatectomy v.s. no3D Intervention: a Prospective Multicenter Randomized Controlled Trial
Brief Title: Artificial Intelligence 3D Augmented Reality Robot-Assisted-Radical- Prostatectomy v.s. no3D Intervention
Acronym: RIDERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Collaborators: San Luigi Gonzaga Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 027-FPO22
Record Dates: First submitted 2024-02-15; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cancer of Prostate
Keywords: 3D AI-AR-RARP; Cancer of Prostate; prostate surgery; Hyper-Accuracy 3D reconstruction (HA3DTM); Riders; computer vision; Robot-assisted; laparoscopic radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized using an Excel® macro in 2 group: 3D and no3D, stratifying them by age, PSA, cT, PSA density, prostate volume, lesion volume, extracapsular extension (ECE), seminal vesicle invasion (SVI), biopsy ISUP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D group (Experimental): in Group 3D, an intrafascial nerve-sparing (NS) technique will be performed on the side of the lesion; contralaterally an intra-, inter- or extra-fascial NS technique will be performed. After removal of the prostate, virtual images of the prostate will be projected into the lodge using AI software and will be displayed thanks to the Tile-Pro. The virtual 3D model will allow identifying the extracapsular extension of the tumor lesion, projected at the level of the preserved neurovascular bundle.
  A first selective excisional biopsy at the level of the suspected ECE on the NVB will be sent for extemporaneous histological examination. Under 3D AR guidance, a second selective biopsy will then be performed on the NVB at the same level as the first, however involving a larger and thicker layer of tissue. the biopsies will be sent for extemporaneous histological examination. In case of positivity, the entire NVB will be removed
  Interventions: Procedure: 3D Robot-assisted laparoscopic radical prostatectomy and pelvic lymphadenectomy
- no3D group (Active Comparator): For the no-3D group, the intra-, inter- or extra-fascial NS technique during robotic prostatectomy will be performed according to the clinical indication.
  At the end of the demolitive phase a selective biopsu was performed in a cognitive fashion accordin with the information provided by MRI images.
  Reconstructive phase was performed according to our previously described total anatomical reconstruction (TAR) technique for both arms.
  Interventions: Procedure: 3D Robot-assisted laparoscopic radical prostatectomy and pelvic lymphadenectomy

INTERVENTIONS:
Procedure: 3D Robot-assisted laparoscopic radical prostatectomy and pelvic lymphadenectomy — The operation is performed using the "Da Vinci HD" robotic system which allows the use of laparoscopic instruments, with greater mobility and the possibility of easier and more precise control of movements in three dimensions. Furthermore, the system allows the surgeon a three-dimensional view of the operating field. The surgery is performed under general anesthesia. Six or more trocars are positioned, into which the instruments operated by the robot or directly by the surgical assistants are inserted.
  Then a radical prostatectomy is performed.

SUMMARY:
This is a prospective randomized multicenter study aimed at comparing 3D AI-AR-RARP vs. no 3D, verifying the impact of this new technology on oncological and functional outcomes after the procedure.

DETAILED DESCRIPTION:
Considering that prostate cancer lesions are not identifiable during surgery, except in the case of extensive and advanced tumors, the surgeon does not have a real-time perception of the location of the tumor. The absence of clear spatial visualization can therefore lead to a positive surgical margin, particularly in tumors in the T3 stage (invasion of the prostatic capsule or seminal vesicles).

Our hypothesis is that with the help of AI 3D AR during surgery, positive surgical margins can be avoided, or at least reduced, while preserving the neurovascular bundles, with a consequent improvement not only in postoperative functional outcomes (continence and potency), but also oncological ones (less biochemical disease recovery (BCR), less need for salvage radiotherapy, lower risk of metastasis).

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the written informed consent and consent to the use of personal data
2. Age > 40 years and male sex
3. Pre-operative MRI performed according to ESUR recommendations and reporting in accordance with PiRads V.2
4. Disease with evidence of bulging or radiological T3 on pre-operative MRI
5. Histological diagnosis of acinar type prostate cancer in the area highlighted on MRI
6. Absence of bulky (>3 cm), bony or visceral retroperitoneal or pelvic lymph node metastatic lesions
7. Patients eligible for radical prostatectomy + pelvic lymphadenectomy
8. ECOG PS 0-1
9. Life expectancy ≥ 5 years
10. Patients motivated to preserve erection and with pre-operative sexual activity with IIEF >17
11. Availability of the patient's pre-operative clinical data
12. Patients must be available to carry out the visits foreseen in the follow-up of the protocol and consent to data collection

Exclusion Criteria:

1. Special histotypes of prostate cancer
2. Patients with PSA > 100 ng/ml at diagnosis
3. Inability to perform MRI (pacemaker wearers, claustrophobia...) or MRI of inadequate quality to obtain the HA3DTM 3D reconstruction
4. Concomitant treatment with other antineoplastic drugs including investigational endocrine therapies
5. Serious uncontrolled concomitant medical condition or disease including active, uncontrolled infections
6. Patients with dementia or psychiatric illness that limit compliance with study requirements or that may prevent understanding and/or signing informed consent.

Ages: 40 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative surgical oncological outcomes | 12 months after surgery
  Verify oncological outcomes in prostate cancer patients with evidence of bulging or extracapsular disease (ECE or rT3) on preoperative MRI, in terms of positive margin rate (PSM) following surgery

SECONDARY OUTCOMES:
Micturition outcomes | 5 years after surgery
  Evaluation of continence recovery rate. Continence was defined as use of 0-1 pads/die. Furthermore 24/h pad test was performed in case of persistence of incontinence to evaluate the different degree of urine losses, and was classified according to ICS definitions.
Sexual function outcomes | 5 years after surgery
  Evaluation of erection recovery in terms of IIEF-5 (International Index of Erectile Function Questionnaire).
Oncological outcomes | 5 years after surgery
  Evaluation of patients' oncological outcomes during the follow up in terms of biochemical recurrence (BCR) and occurrence of local/distant recurrence detected with different imaging techniques during the FU according to clinical indication

OTHER OUTCOMES:
Verify the potential application of AI | 12 months after surgery
  Verify the potential application of AI as an alert system during surgery in order to reduce the rate of possible intraoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Checcucci, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo
Locations (2):
- Italy (2):
  - Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin
  - AOU san Luigi Gonzaga, Orbassano, Turin